CLINICAL TRIAL: NCT01925456
Title: Validation of Instruments for Pragmatic Clinical Trials for Overatcive Bladder
Brief Title: Validation of Instruments for Pragmatic Clinical Trials for Overactive Bladder
Acronym: PfizerOABLUT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 813672
Record Dates: First submitted 2013-08-06; First posted 2013-08-19 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2011-06

CONDITIONS: Overactive Bladder
Keywords: urge urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Toviaz (Other): Patients willingness to take Toviaz 4mg and 8mg
  Interventions: Drug: Toviaz

INTERVENTIONS:
Drug: Toviaz — Means of effectiveness, adherence, and utility instruments over time will be examined to evaluate whether changes are linear from baseline to 8 weeks and 3 months. We will demonstrate the validity and responsiveness of pragmatic instruments against existing established measures (Table 3).
  Other Names: Toviaz4mg and 8mg

SUMMARY:
A. Objectives & Hypothesis Overactive bladder (OAB) affects over 10 million adults in the United States and each year substantial costs are incurred from private and public funds to test the efficacy of new and existing drugs for OAB.14 However, effectiveness and adherence data from traditional clinical trials are not generalizable to clinical practice.3, 4 In an era of limited resources and competing demands, it is essential that cost-effectiveness data from clinical trials be generalizable to the clinical world. Pragmatic clinical trials measure the effectiveness of treatments in real clinical practice, and in the full spectrum of patients that require treatment.5 Pragmatic trials require patient reported outcomes that are valid but have low patient burden.5 The conduct of pragmatic clinical trials for OAB has been limited by a lack of instruments that have demonstrable validity and reliability in the typical clinical setting Pill counts, used to measure primary outcomes in most traditional trials, are burdensome in the clinical setting.1610 The optimal instrument for measuring utility scores, general quality of life scores for cost-effectiveness analyses for OAB, is also not known.

Although poor adherence carries the potential for continued suffering for patients and wasted health care resources, there is a lack of data on the clinical and economic impact of poor adherence to treatment for OAB in real-world clinical practice. We have published preliminary data that underscores the role of adherence and utilities in the treatment of OAB. 3 Our hypothesis is that effectiveness, adherence, and utility preference scores can be measured using pragmatic patient reported instruments and that poor adherence is associated with lower effectiveness and quality of life in adults with OAB in a clinical setting. Specifically, the overriding goal of this proposal is to validate pragmatic instruments to measure effectiveness, adherence and utility preference scores and obtain preliminary data on the effect of adherence and quality of life in adults undergoing treatment for overactive bladder in a clinical setting.

DETAILED DESCRIPTION:
Specific Aim 1: To determine the validity and responsiveness of pragmatic patient reported outcome instruments to measure clinical effectiveness, adherence and utility preference scores in adults undergoing treatment with anti-cholinergic medications for overactive bladder. We will perform a prospective cohort study of adults with OAB undergoing treatment with anti-cholinergic medication. We will compare improvement in urinary symptoms (clinical effectiveness), adherence, and change in utility preference scores from baseline to 3 months of treatment using new and existing 'gold standard' instruments. The results will be informative as to which, if any of these pragmatic instruments, is useful for measuring effectiveness, adherence, and utility preference scores in the 'real world' clinical setting.

Specific Aim 2: To use the newly validated pragmatic instruments to measure the impact of adherence on clinical effectiveness and health related quality of life in a real world clinical setting in adults undergoing treatment with anti-cholinergic medications for overactive bladder. The impact of adherence on clinical effectiveness and health related quality of life will be measured through comparisons in adults with high and low adherence to anti-cholinergic medication. This aim will corroborate the findings of aim 1 and establish if pragmatic instruments are useful in measuring outcomes of effectiveness, adherence and utility preference scores. These results will also provide preliminary data on the effectiveness of anti-cholinergic medication and the impact of adherence on clinical effectiveness and quality of life in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

1. urinary urgency for at least 3 months.
2. Subjects must have mean of ≥ 8 voids per 24 hours
3. and ≥ 1 urgency episode per 24 hours and a rating of at least moderate bother on the single item
4. Patient Perception of Bladder Condition.

Exclusion Criteria:

1. < 18 years
2. predominant stress incontinence as measured by the validated 3-Incontinence Questionnaire
3. current/recent use (≤6 m) or contra-indication to anti-cholinergic medication for OAB
4. severe voiding difficulties in the judgment of the investigator
5. men on unstable use of alpha blockers/5-alpha reductase inhibitors
6. severe neurologic disease
7. anti-incontinence or prolapse surgery
8. pregnancy ≤6 months
9. pelvic neuromodulation other lower urinary tract disorder such as calculus, urethral diverticulum, current or recurrent urinary tract infections.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Clinical effectiveness The primary outcome for clinical effectiveness will be patient reported improvement in urinary urgency at 3 months compared to before start of treatment. On two pragmatic instruments, QVD and OAB-q clinical effectiveness will be | 2.5 YEARS
  QVD-Questionnaire Based Voiding Diary

CONTACTS AND LOCATIONS:
Overall Officials: Lily A Arya, MS, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania 3400 Spruce Street-1000 Courtyard, Philadelphia, Pennsylvania, United States